CLINICAL TRIAL: NCT04000867
Title: Treatment for Foot Pain Caused by Diabetic Neuropathy Using Recurrent TransCutaneous Magnetic Stimulation (TCMS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: ZyGood LLC (Industry)
Collaborators: University of Maryland (Other); Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TCMS for DN
Record Dates: First submitted 2019-06-19; First posted 2019-06-27 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Diabetic Peripheral Neuropathy
Keywords: diabetic foot pain; diabetic foot neuropathy; diabetic foot numbness

STUDY DESIGN:
Intervention Model Description: Multi-site double blinded randomized control clinical trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: 20 patients given the choice of 1 out of 20 envelopes they pick, 10 will be randomized to either the real TCMS treatment arm or 10 to the sham treatment arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- real TCMS treatment (Active Comparator): Subjects with DN located in their bilateral feet that have been previously identified and have a graded average baseline score of at least 5 in each foot will receive either TCMS treatment or Sham treatment on clinic day-1 according to the contents of a sealed opaque envelope corresponding to the subject's number in the series and opened immediately before treatment on day 1. (Our statistician will have generated these envelopes and their contents in advance.) Subjects and staff evaluating the subject's response will remain blinded to treatment assignment; only the staff member setting the treatment mode will know whether it is active or sham.
  Interventions: Device: Transcutaneous Magnetic Stimulation (TCMS)
- Sham TCMS treatment (Sham Comparator): Patients in the sham treatment group, will use the same device. The device will be switched into sham mode by the clinician by pressing a small, non-descript button on the backside of the pulse generator. The treatment device in sham mode will produce a clicking sound once every 6 seconds like the TCMS treatment mode, but no magnetic pulses will be output.
  Interventions: Device: Transcutaneous Magnetic Stimulation (TCMS)

INTERVENTIONS:
Device: Transcutaneous Magnetic Stimulation (TCMS) — The study will evaluate whether an experimental medical device that emits a series of brief, intense magnetic pulse called TCMS will relieve foot pain from Diabetic Neuropathy (DN) when compared to the same device giving a sham treatment without magnetic pulses. Participants will be blindly randomized into either the TCMS treatment group or the sham treatment group according to the number 1-20 that they draw. This is necessary to further investigate this TCMS treatment and to determine how to obtain statistically significant data as to whether this therapy reduces the foot pain caused by diabetic neuropathy.

SUMMARY:
The study will evaluate whether an experimental medical device that emits a series of brief, intense magnetic pulse will relieve foot pain from Diabetic Neuropathy (DN) if used weekly for a month

DETAILED DESCRIPTION:
The study will evaluate whether an experimental medical device that emits a series of brief, intense magnetic pulse will relieve foot pain from Diabetic Neuropathy (DN) if used weekly for a month The United States Food and Drug Administration (FDA) has approved a similar device for treatment of migraine headaches, but this type of device has not been studied for the treatment of DN. No significant adverse reactions or side effects have been reported from the use of magnetic stimulation for the headache treatment or for the treatment of foot pain for about 20 patients. Some patients who have migraine headaches or foot pain have excellent pain relief with the magnetic treatment even if they did not get pain relief using medications.

The initial safety and feasibility study did show it was both safe and effective but short term with most benefits wearing off after 1 week. Additionally in the initial study no placebo comparisons were made, therefore this study will consist of 20-blinded randomized patients. 10 will receive the TCMS treatment weekly and 10 will receive a sham treatment weekly both for 1 month.

Investigators believe that using the device weekly will relieve the foot pain caused by diabetic neuropathy over the course on 1 month compared with those receiving the sham treatment.

And to prove this hypothesis investigators will treat 10-blinded patients in the TCMS treatment group, they will be receiving active treatment as follows:

50 pulses to the sole of the patient's left (L) foot by placing the foot on top of the device with the heel touching the heel stop (the rear position)

Then followed by another 50 pulses to sole of the patient's L foot by either:

Moving the foot forward so the toes touch the toe stop (the forward position) or By placing the patients' foot under the pulsing deck (the under-deck position)

This procedure will then be repeated for the right (R) foot

10-blinded patients in the sham treatment group will use the same device. However, device will be switched into sham mode by the only un-blinded clinician in the study by pressing a small, non-descript button on the backside of the pulse generator. The treatment device in sham mode will produce a clicking sound once every 6 seconds like the TCMS treatment mode, but no magnetic pulses will be output.

Patients will receive the sham treatment the same as the TCMS treatment group, as described above and both groups will be completing a daily diary to rate and evaluate their pain and their quality of life for the month they participate in the study.

One side effect of this treatment may be some muscular jerking of the foot or the toes during the application of the magnetic pulses. This jerking will last only during the treatment and will not be painful or harmful.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years of age.
2. Pain duration of more than one month.
3. Pain occurs daily.
4. Chronic DN associated bilateral foot pain and is not explained by a central anatomic nerve compression and can clearly be correlated with that patient's history of diabetes.
5. Average Pain intensity ≥ 5 in each foot for at least 3 days at the time of enrollment.

Exclusion Criteria:

1. Life expectancy ≤ 6 months.
2. Oral pain medication doses or active ingredient has changed significantly* in the prior 2 weeks.
3. Inability to walk at least 10 steps (with or without a cane/walker) before and after having to sit in a chair.
4. Another pain condition that might confound results (e.g., neuropathy from cancer chemotherapy, plantar fasciitis or arthritis of ankle and foot)
5. Inability to undergo study assessments or complete questionnaires independently.
6. Active psychological co-morbidities (i.e., uncontrolled schizophrenia).
7. Currently using an opioid medication for the treatment of foot pain**.
8. Pregnancy
9. Inability to have MRI
10. Metal hardware and/or fragments in feet and ankles
11. Implanted pacemaker or a defibrillator, unless the device is considered MRI safe

    * A significant change for this study is defined as a 20% increase or decrease in dosing of the patient's medication dose and/or or a change in the medication class (adding or removing other types of medicines used to treat pain).

      * This exclusion is restricted to opioids, benzodiazepines and psychotropic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
Overall Pain reduction | 28 day +/- 2 days
  The primary endpoint will be defined as achieving at least reduction in average pain score from 0-10 (0 being no pain and 10 being the worst pain imaginable) )versus the sham control using pre-study average baseline for each subject as a covariate by a repeated measures analysis of pain scores through 28 days.

SECONDARY OUTCOMES:
Pain reduction with in the first week | 1 week
  Secondary endpoints will include a responder analysis in which the percentage of subjects between the sham and test groups that achieve the minimum clinically important pain reduction of 2 or more points from the scale described above within the first week of treatment.
Improved Activities of daily living | 28 days +/- 2 days
  Secondary endpoints will also include improved quality of life (ie, 1-Did the level of your pain interfere with your daily activities at home or work? 2-Did the level of your pain interfere with your social or recreational activities? 3-Did the level of your pain interfere with your sleep?) the responses as guided by the PROMIS questions ( answered as one of 5 choices Not at All A little bit Somewhat Quite a bit Very Much) included in the pre and post questionnaires and the home assessment diary booklet.

CONTACTS AND LOCATIONS:
Overall Officials: Kashif Munir, MD, Principal Investigator — University of Maryland; Ejaz Shamim, MD, Principal Investigator — Kaiser Permanente

IPD SHARING:
Plan to Share IPD: Undecided
not yet decided